CLINICAL TRIAL: NCT06133140
Title: Continuous Ward Monitoring With the GE Portrait Mobile Monitoring Solution: the COSMOS Trial
Acronym: COSMOS
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 24-009
Record Dates: First submitted 2023-11-01; First posted 2023-11-15 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Complications
Keywords: Postoperative; Anesthesia; Vital signs
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Blinded monitoring: Continuous postoperative vital sign monitoring blinded to clinicians and investigators.
  Interventions: Device: Blinded postoperative vital sign monitoring
- Unblinded monitoring: Continuous postoperative vital sign monitoring unblinded to clinicians and investigators.
  Interventions: Device: Unblinded postoperative vital sign monitoring

INTERVENTIONS:
Device: Unblinded postoperative vital sign monitoring — Unblinded postoperative GE Portrait monitoring
  Other Names: Unblinded group
  Groups: Unblinded monitoring
Device: Blinded postoperative vital sign monitoring — Blinded postoperative GE Portrait monitoring
  Other Names: Blinded group
  Groups: Blinded monitoring

SUMMARY:
The investigators plan to determine whether unblinded continuous ward monitoring with the GE Portrait Mobile Monitoring Solution and nursing alerts reduces vital sign abnormalities in patients recovering from major noncardiac surgery.

DETAILED DESCRIPTION:
Primary Aim. Determine whether unblinded continuous ward monitoring with the GE Portrait Mobile Monitoring Solution and nursing alerts reduces vital sign abnormalities in patients recovering from major noncardiac surgery.

Primary hypothesis. Unblinded continuous ward monitoring and nurse alerts reduces vital sign abnormalities during the initial 48 postoperative hours after major non-cardiac surgery while patients remain hospitalized.

Secondary Aim. Determine whether continuous ward saturation, ventilation, and pulse rate monitoring reduces a composite of substantive respiratory and cardiovascular interventions.

Secondary hypothesis. Unblinded continuous ward monitoring increases a composite of clinical interventions for desaturation, hypoventilation, tachypnea, tachycardia, and bradycardia within 48 hours after major non-cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Are expected to be admitted to one of the wards equipped with the GE Portrait Mobile Monitoring Solution;
2. Are ≥18 years old;
3. Are designated American Society of Anesthesiologists physical status 1-4;
4. Are scheduled for major noncardiac surgery lasting at least 1.5 hours;
5. Are expected to remain hospitalized at least one postoperative night;
6. Are expected to have general or neuraxial anesthesia.

Exclusion Criteria:

1. Have language, vision, or hearing impairments that might compromise continuous monitoring;
2. Are designated Do Not Resuscitate, hospice, or receiving end of life care;
3. Are expected to have telemetry monitoring;
4. Have previously participated in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are older than 18 years of age. Patients have a ASA status 1-4. The patients whom had a major noncardiac surgery lasting at least 1.5 hours and are expected to remain hospitalized at least two postoperative nights, and are being admitted to a ward equipped with the GE Portrait Mobile Monitor.
Sampling Method: Probability Sample
Enrollment: 227 (Actual)
Dates: Start 2024-02-14 (Actual); Primary Completion 2026-01-01 (Actual); Study Completion 2026-01-06 (Actual)

PRIMARY OUTCOMES:
Hypoxemia | 48 postoperative hours.
  Area of oxygen saturation defined as SpO2 ≤85%.
Inadequate or excessive ventilation | 48 postoperative hours.
  Area of inadequate or excessive ventilation defined as respiratory rate ≤4/min or ≥30/min.
Bradycardia and tachycardia | 48 postoperative hours.
  Area of inadequate or excessive heart rate defined as ≤40/min or ≥130/min.

SECONDARY OUTCOMES:
The fraction of patients who have a composite of interventions potentially related to postoperative vital sign abnormalities. | 48 postoperative hours.
  Determine whether continuous ward saturation, ventilation, and pulse rate monitoring reduces substantive respiratory and cardiovascular interventions. Each intervention will be considered dichotomously (occurred or not), and together constitute a composite outcome:
  * Supplemental oxygen (or substantive dose escalation as indicated by a new administration method) excluding oxygen that patients are already using when they arrive on the ward;
  * New-onset inhaled drugs (e.g., steroids, bronchodilators);
  * Naloxone or flumazenil administration;
  * Non-invasive ventilatory support including bag & mask ventilation, but excluding use of home CPAP and similar devices;
  * Bolus fluid administration (e.g., >500 ml);
  * Drug treatments for bradycardia (e.g., new onset atropine or glycopyrrolate) and discontinuing drugs that promote bradycardia such as beta blockers;
  * Drug treatment for tachycardia (e.g., new onset beta blockers and calcium channel blockers).

CONTACTS AND LOCATIONS:
Overall Officials: Ryu Komatsu, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared collaboratively upon approval of the Steering Committee and appropriate data-use agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: One year after publication of main paper.
Access Criteria: Contact PI.